CLINICAL TRIAL: NCT01034306
Title: A Phase IIB Study of the Efficacy and Safety of Daily CF101 in Patients With Active Rheumatoid Arthritis and Elevated Baseline Expression Levels of Peripheral Blood Mononuclear Cell A3 Adenosine Receptors
Brief Title: Oral CF101 Tablets Treatment in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF101-204RA
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — CF101; N(6)-(3-iodobenzyl)-5'-N-methylcarboxamidoadenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CF101 1 mg (Experimental): piclidenoson (CF101) 1 mg tablet oral, Q12h for 12 weeks
  Interventions: Drug: CF101
- Placebo (Placebo Comparator): placebo tablet to match the active, oral dosage, Q12h for 12 weeks
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: CF101 — orally q12h
  Other Names: IB-MECA
  Arms: CF101 1 mg
Drug: Placebo control — orally q12 hours
  Other Names: Inactive pill
  Arms: Placebo

SUMMARY:
This trial will test the hypothesis that the administration of CF101, a novel anti-inflammatory agent, to patients with rheumatoid arthritis and high A3AR expression at baseline will relieve signs and symptoms of the disease.

DETAILED DESCRIPTION:
This will be a multi-center, randomized, double-blind, parallel-group, placebo-controlled, study in which patients with active RA and high A3AR expression at baseline will be randomized to the addition of either CF101 1.0 mg or placebo given orally q12h for 12 weeks. Screening examinations will occur within 1 month prior to dosing. Washout of other disease-modifying antirheumatic drugs (DMARDs), including biological agents, will occur prior to dosing; if washout is necessary, patients must re-qualify for inclusion following the washout. Doses of nonsteroidal anti-inflammatory drugs (NSAIDS) and corticosteroids must be stable for >=1 month prior to dosing and remain so during protocol participation. Disease activity will be assessed using swollen and tender joint counts, physician and patient global assessments (by visual analog scale, VAS), patient reported pain (by VAS), a Health Assessment Questionnaire (HAQ) Disability Index (DI), Westergren erythrocyte sedimentation rate (ESR, Screening, Weeks 0 and12), and C-reactive protein (CRP) levels. Assessments will take place at Screening, Baseline (Week 0), and at Weeks 2, 4, 8, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 18-75 years
* Meet the criteria of the American College of Rheumatology for RA (Arnett FC et al. Arthritis Rheum 1988;31:315-324, Appendix 1)
* Not bed- or wheelchair-bound
* Active RA, as indicated by the presence of (a) >=6 swollen joints (28 joint count); AND (b) >=6 tender joints (28 joint count); AND either: (c) Westergren ESR of >=28 mm/hour; OR (d) CRP level above the upper limit of normal for the central reference laboratory
* Elevated PBMC A3AR expression level, defined as >= 1.5-fold over a predetermined normal population standard, following the appropriate DMARD/biologic washout period (see Exclusion Criteria) but within 2 weeks of beginning dosing
* If taking a nonsteroidal anti-inflammatory agent (NSAID), dose has been stable for at least 1 month prior to the A3AR Qualification Visit, and will remain unchanged during protocol participation
* If taking an oral corticosteroid, dose is <=10 mg/day prednisone or equivalent, has been stable for at least 1 month prior to the A3AR Qualification Visit, and will remain unchanged during protocol participation
* In the Investigator's opinion, the ability to understand the nature of the study and any hazards of participation, and to communicate satisfactorily with the Investigator and to participate in, and to comply with, the requirements of the entire protocol
* Negative screening serum pregnancy test for female patients of childbearing potential
* Females of childbearing potential must utilize, throughout the course of the trial, 2 methods of contraception deemed adequate by the Investigator (for example, oral contraceptive pills plus a barrier method)
* All aspects of the protocol explained and written informed consent obtained

Exclusion Criteria:

* Receipt of any of the following for at least a 1 month washout period prior to the A3AR Qualification Visit: methotrexate, sulfasalazine, oral or injectable gold, azathioprine, minocycline, penicillamine, anakinra
* Receipt of etanercept for at least a 6 week washout period prior to the A3AR Qualification Visit
* Receipt of chloroquine, hydroxychloroquine, cyclosporine, infliximab, golimumab or adalimumab for at least a 2 month washout period prior to the A3AR Qualification Visit
* Receipt of leflunomide for at least a 2 month washout period prior to the A3AR Qualification Visit, unless patient has undergone cholestyramine washout at least 1 month prior to testing
* Receipt of cyclophosphamide for at least a 6 month period prior to the A3AR Qualification Visit
* Receipt of rituximab at any previous time
* Previous failure to respond to methotrexate or any anti-rheumatic biological agent
* Participation in a previous trial CF101 trial
* Use of oral corticosteroids >10 mg of prednisone, or equivalent, per day
* Change in NSAID dose level for 1 month prior to the A3AR Qualification Visit
* Change in oral corticosteroid dose level during the 1 month prior to the A3AR Qualification Visit
* Receipt of parenteral or intra-articular corticosteroids during the 1 month prior to the A3AR Qualification Visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2010-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Director — BioStrategics Consulting Ltd
Locations (5):
- Bulgaria (4):
  - Multiprofile Hospital for Active Treatment, Sofia
  - Diagnostic Consultative Center Sofia, Sofia
  - Military Medical Academy, Sofia
  - UMHAT "Sveti Ivan Rilski", Rheumatoloty Clinic, Sofia
- Barzilai Medical Center, Ashkelon, Israel

REFERENCES:
- See also: Sponsor — http://www.canfite.co.il

RESULTS

PARTICIPANT FLOW:
Groups:
- CF101 1mg: CF101 1mg q12 for 12 weeks
- Placebo: Matching placebo q12 for 12 weeks
Period: Overall Study
Arm/Group | CF101 1mg | Placebo
Started | 42 | 37
Completed | 37 | 34
Not Completed | 5 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — hospitalized and decided to stop | 1 | 0
Not completed — Noncomplience | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CF101 1mg | Placebo | Total
Number analyzed (Participants) | 42 | 37 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (9.87) | 61.7 (6.89) | 59 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving an American College of Rheumatology 20 (ACR20) Response (20% Improvement)
Description: ACR20 Response is defined as a 20% improvement from baseline in disease:
  1. >20% improvement in tender joint count (TJC), and
  2. >20% improvement in swollen joint count (SJC), and
  3. >20% improvement in at least 3 of following 5:
     1. Physician global assessment (PGA),
     2. Patient global assessment (PAGA),
     3. Patient pain assessment (PPA),
     4. Patient's assessment of physical function using Health Assessment Questionnaire (HAQ), and
     5. Most improved response of ESR and CRP
Time Frame: 12 weeks
Population: ITT population, all-cause dropouts considered non-responders
Measure: Count of Participants; unit: Participants
Arm/Group | CF101 1mg | Placebo
Number analyzed (Participants) | 42 | 37
Participants | 18 | 8
Statistical Analysis 1: Comparison: CF101 1mg vs Placebo; Test type: Superiority; p = 0.0352, t-test, 2 sided — normal approximation to the binomial test

2. Secondary Outcome: Number of Subjects Achieving an ACR50 Response (50% Improvement)
Description: ACR50 Response is defined as a 50% improvement from baseline in disease:
  1. >50% improvement in TJC, and
  2. >50% improvement in SJC, and
  3. >50% improvement in at least 3 of following 5:
     1. Physician global assessment (PGA),
     2. Patient global assessment (PAGA),
     3. Patient pain assessment (PPA),
     4. Patient's assessment of physical function using Health Assessment Questionnaire (HAQ), and
     5. Most improved response of ESR and CRP
Time Frame: 12 weeks
Population: ITT population, all-cause dropouts considered non-responders
Measure: Count of Participants; unit: Participants
Arm/Group | CF101 1mg | Placebo
Number analyzed (Participants) | 37 | 32
Participants | 7 | 3
Statistical Analysis 1: Comparison: CF101 1mg vs Placebo; Test type: Superiority; p = .2472, t-test, 2 sided

3. Secondary Outcome: Number of Subjects Achieving an ACR70 Response (70% Improvement)
Description: ACR70 Response is defined as a 70% improvement from baseline in disease:
  1. >70% improvement in TJC, and
  2. >70% improvement in SJC, and
  3. >70% improvement in at least 3 of following 5:
     1. Physician global assessment (PGA),
     2. Patient global assessment (PAGA),
     3. Patient pain assessment (PPA),
     4. Patient's assessment of physical function using Health Assessment Questionnaire (HAQ), and
     5. Most improved response of ESR and CRP
Time Frame: 12 weeks
Population: ITT population, all-cause dropouts considered non-responders
Measure: Count of Participants; unit: Participants
Arm/Group | CF101 1mg | Placebo
Number analyzed (Participants) | 37 | 32
Participants | 4 | 1
Statistical Analysis 1: Comparison: CF101 1mg vs Placebo; Test type: Superiority; p = 0.1972, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | CF101 1mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/42 | 1/37
Other Adverse Events (participants affected / at risk) | 0/42 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CF101 1mg (N=42) | Placebo (N=37)
Pyoderma (Infections and infestations) | 1 | 0 — Pyoderma
atrial fibrillation with uncontrolled ventricular response (Cardiac disorders) | 0 | 1 — atrial fibrillation with uncontrolled ventricular response

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No